CLINICAL TRIAL: NCT01334697
Title: Phase I, Randomized, Multicenter, Double-blind, Single Dose, Dose-Escalation, Placebo-Controlled, Parallel Group Clinical Trial to Investigate the Safety, Tolerability and Pharmacokinetics of Intravenous Administration of Cardiotrophin-1 (CT-1)in Healthy Volunteers
Brief Title: Clinical Trial to Assess the Safety, Tolerability and Pharmacokinetics of Cardiotrophin-1 in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Digna Biotech S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: CT1-HEPT-01, 2010-022929-15
Record Dates: First submitted 2011-04-05; First posted 2011-04-13 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Healthy
Keywords: Cardiotrophin-1; CT-1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cardiotrophin-1 (Experimental)
  Interventions: Drug: recombinant human cardiotrophin-1
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: recombinant human cardiotrophin-1 — Single dose intravenous administration
  Arms: Cardiotrophin-1
Other: Placebo — Single dose intravenous administration
  Arms: Placebo

SUMMARY:
The general aim of the study is to determinate safety, tolerability and early pharmacokinetics of cardiotrophin.1 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, between the ages of 18 and 55.
* Healthy condition (no suffering from known acute or chronic disease)
* No clinically important abnormal physical or laboratory findings at the screening examination.
* Normal or clinically acceptable ECG.
* Normal blood pressure (systolic: 90-140 mmHg; diastolic: 50-90 mmHg) and heart rate (40-100 bpm).
* Body Mass Index of 19.0-29.0 (kg/m2).
* Ability to communicate well with the investigator and to comply with the requirements of the entire study.
* Willingness to give written informed consent (prior to any study-related procedures being performed) and to be able to adhere to the study restrictions and examination schedule.
* For female subjects with childbearing potential: use of a known highly effective method of birth control, defined as those which results in a low failure rate: i.e. less 1% per year, (contraceptive pills, intrauterine contraceptive device, implants, vasectomized partner or sexual abstinence), for at least three consecutive months prior to the study, during the study and one month after the end of the study.
* For male subjects with partners of child bearing potential: use of appropriate contraceptive methods (vasectomy, condoms or sexual abstinence), for at least the study period and one month after the end of the study.

Exclusion Criteria:

* Administration of any investigational drug in the period within three months prior to informed consent.
* Use of any prescription medication during the period 0 to 30 days or over-the-counter medication during the 0 to 5 days before entry to the study.
* Donation or loss of greater than 400 ml of blood in the period 0 to 12 weeks before entry to the study.
* Serious adverse reaction or hypersensitivity to any drug.
* Inability to communicate or co-operate with the investigator because of a language problem, poor mental development or impaired cerebral function.
* History of drug dependence (except tobacco) or psychiatric illness within the past 2 years.
* Consumption of alcohol within 24 hours prior to dose administration.
* Presence of pain incurred by unknown causes.
* Pregnancy or nursing.
* Positive urine drug screen for drugs with a high potential for abuse and low persistence in the urine.
* Inability to refrain from smoking during study days.
* Any other condition which, in the opinion of the investigators, is likely to interfere with the successful collection of the measures required for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events as a Measure of Safety and Tolerability | single dose administration (baseline) and 1 post-treatment follow up week
  Evaluate the tolerability and safety of single dose intravenous administration

SECONDARY OUTCOMES:
Pharmacokinetic and Pharmacodynamic parameters | single adminsitration (baseline) and 1 week of follow up
  Obtain pharmacokinetic parameters before and after CT-1 single dose administration.
  Analyze surrogated biological markers associated with CT-1 administration

CONTACTS AND LOCATIONS:
Overall Officials: Belén Sádaba, MD, Principal Investigator — Clínica Universidad de Pamplona
Locations (2):
- Spain (2):
  - Hosp. Universitario Puerta de Hierro de Majadahonda, Madrid
  - Clínica Universidad de Navarra, Pamplona

REFERENCES:
- See also: Treatment of murine fulminant hepatitis with genetically engineered endothelial progenitor cells. — http://www.ncbi.nlm.nih.gov/pubmed/21334399
- See also: [Obesity, inflammation and insulin resistance: role of gp 130 receptor ligands]. — http://www.ncbi.nlm.nih.gov/pubmed/18953360